CLINICAL TRIAL: NCT04188678
Title: REBOUND: REsiliency in Older Adults UNDergoing BOne Marrow Transplant - A Pilot Study of Resiliency Measures in Older Patients Undergoing Allogeneic Blood and Marrow Transplant
Brief Title: Resiliency in Older Adults Undergoing Bone Marrow Transplant
Acronym: REBOUND
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: J1849; UH2AG056933 (NIH); IRB00165139 (Other: Johns Hopkins School of Medicine)
Record Dates: First submitted 2019-11-26; First posted 2019-12-06 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Leukemia; Lymphoma; Blood Cancer; Myelodysplastic Syndrome; Acute Myelogenous Leukemia; Non-Hodgkins Lymphoma
Keywords: Allogeneic blood and marrow transplantation (alloBMT); Resiliency; REBOUND; over age 60
MeSH Terms: conditions — Leukemia; Lymphoma; Hematologic Neoplasms; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin | interventions — Bone Marrow Transplantation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interventional Arm- Bone Marrow Transplant: Study visits will include the performance of assessments prior to the start of conditioning chemotherapy and at 1 month and 6 months post-BMT. Assessments include:
  1. Physical function assessments
  2. questionnaires about general health and current health compared to health one year ago
  3. assessments that measure cognition, attention and memory
  4. assessments regarding personality and psychological and social stressors
  5. Physiological measures including
     * blood tests- 160 mL of blood during evaluations, and 90mL of blood at the day 180 visit.
     * bone marrow aspirate collected during standard of care bone marrow biopsies pre-transplant and at day 180
     * Saliva collections pre-transplant
     * ACTH Stimulation Test
     * Oral Glucose Tolerance Test
     * Holter Monitor- to record hear rate variability
     * MRI pre-transplant and at Day 180 in a subset of 10 subjects
  Interventions: Other: Bone Marrow Transplant (BMT)

INTERVENTIONS:
Other: Bone Marrow Transplant (BMT) — Bone marrow transplantation will be conducted according to the investigators' institution's standard of care, or else according to research protocol (if applicable).Study visits that include the performance of assessments will occur prior to the start of conditioning chemotherapy and at 1 month and 6 months post-BMT. All dates are +/- 7 days. The initial study visit will take place during standard of care pre-transplant evaluations, which typically span 3-4 days. The post-BMT visits will take place before or after regularly-scheduled BMT follow up.

SUMMARY:
The objective of this research is to measure certain indicators of resiliency to better understand which participants who are over 60 years old will respond more positively to bone marrow transplant. This research is being done to determine if there are traits that make recipients more likely to bounce back following allogeneic bone marrow transplant (BMT).

DETAILED DESCRIPTION:
Allogeneic blood and marrow transplantation (alloBMT) is the only potentially curative therapy for many forms of leukemia, lymphoma, and other hematologic malignancies. As with many forms of cancer, many of the most common indications for alloBMT disproportionally affect older people. Although treatments have improved for older adults undergoing therapies for these diseases, the outcomes are variable and there is little biological knowledge to help identify specific factors that would predict why some people do well with treatment and others develop functional and cognitive decline and other adverse health outcomes.

Data specific to patients older than 60 who have undergone alloBMT are sparse even though the 1 year non-relapse mortality rate in patients older than age 50 at Johns Hopkins is 12%. In none of these studies have geriatric assessment measures in domains such as cognition and function been evaluated. Given the low incidence of non-relapse mortality in the investigators' older patients, the investigators have a unique opportunity to study the factors that influence not only mortality but function after hematopoietic stem cell transplantation. The investigators aim to be able to counsel patients more specifically about likely outcomes after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing allogeneic bone marrow transplant at Johns Hopkins Hospital, the indication for which is a hematologic malignancy
* Age ≥60 years
* Ability to walk without human assistance
* Enrollment in concomitant clinical research is permitted but not required
* English-speaking
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Unwillingness or inability to return at 6 months after transplantation for repeated evaluation
* Non-English-speaking

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 60 who have undergone alloBMT
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Physical Performance as assessed by Short Physical Performance Battery (SPPB) | Pre-BMT, Day 30 and Day 180 post transplant
  5 measured criteria: unintentional weight loss, exhaustion, low energy expenditure, low grip strength, and slowed waking speed. Scores of 3, 4 and 5 are consistent with frailty, scores of 1 and 2 are consistent with pre-frailty status, and a score of 0 is consistent with a robust or resilient status.
Change in ability to perform activities of daily living as assessed by Instrumental Activities of Daily Living questionnaire | Pre-BMT, Day 30 and Day 180 post transplant
  questions about ability to perform activities of daily living (IADL). Scored low functioning (0) to high functioning (8).
Change in upper extremity function as assessed by accelerometry | 7 consecutive days pre-BMT, at Day 30 and at Day 180
  device worn on wrist for a 24hr period that measures physical activity and sedentary activity. Higher scores= more active.
Change in catecholamines levels as assessed in overnight urine collection samples | Pre-BMT, Day 30 and Day 180 post transplant
  Changes in catecholamines level will be assessed in overnight urine collection samples. Levels fluctuate. Analysis will use the Johns Hopkins University (JHU) normal reference range for an adult is Metanephrine (normotensive):45-290 μg/24 hours. Metanephrine (hypertensive): 35-460 μg/24 hours .
Change in Frailty as assessed by the Frailty Phenotype instrument | Pre-BMT, Day 30 and Day 180 post transplant
  Frailty Phenotype instrument is used to measure participants' walking speed and grip strength, includes questions about exhaustion, physical activity, weight loss. Higher scores indicate better functional state.
Change in Pittsburgh Fatigability Scale for Older Adults score | Pre-BMT, Day 30 and Day 180 post transplant
  self-report tool that normalizes activities in terms of intensity and duration (PFS) this has a range of 0-50 with higher scores indicating greater physical fatigability.
Change in Borg Rating of Perceived Exertion Scale score | Pre-BMT, Day 30 and Day 180 post transplant
  scale will be used immediately after a slow-paced 5-minute treadmill walk to assess fatigability (RPE). Higher score indicates higher perceived exertion.
Change in medical history and diseases/conditions self reporting | Pre-BMT and Day 180 post transplant
  Questionnaire of past medical history as reported by a subject. This questionnaire does not have a score.
Change in health behaviors as assessed by a questionnaire | Pre-BMT and Day 180 post transplant
  This assessment is of self determined overall health as reported by a participant, it has no score.
Change in reporting of patients traumas as assessed by the Hospitalizations, Surgeries, and Falls Questionnaire | Pre-BMT and Day 180 post transplant
  Questionnaire includes items on hospitalizations, surgeries, and falls. it has no score.
Change in pain reporting as assessed by the Pain Assessment Questionnaire | Pre-BMT and Day 180 post transplant
  questions on overall bodily pain intensity/frequency and pain-related function/interference. Higher scores equal more pain.
Change in anxiety reporting as assessed by the anxiety questionnaire | Pre-BMT and Day 180 post transplant
  Questions to assess the presence and severity of anxiety; higher scores = more anxiety.
Change in trauma reporting as assessed by the trauma questionnaire | Pre-BMT and Day 180 post transplant
  Questions to assess a participants reporting of any past experiences of several kinds of trauma. It has no score.
Change in cognitive function as assessed by Modified Mini-Mental State Examination | Pre-BMT, Day 30, Day 56 and Day 180 post transplant
  measure of global cognitive function (range 0-100). A score of 100 represents total cognitive function according to 3MS.
Change in cognitive ability as assessed by the Montreal Cognitive Assessment | Pre-BMT, Day 30, Day 56 and Day 180 post transplant
  measures global cognitive function (MoCA). Scores range between 0 and 30. A score of 26 or over is considered to be normal.
Change in cognitive function as assessed by the Digit Symbol Substitution Test (DSST) | Pre-BMT, Day 30, Day 56 and Day 180 post transplant
  participant fill in a series of symbols correctly coded within 90 seconds. The higher the score, the better the participant's performance.
Change in ability to cope with life challenges as assessed by the Coping Self-Efficacy Scale | Pre-BMT and Day 180 post transplant
  11-point Likert scale measures perceived ability to cope effectively with life. Scale is 0-10 with 10 = best ability to cope and 0 = no ability to cope.
Change in sense of well-being as assessed by the Subscale of Ryff Psychological Well-being Scale | Pre-BMT and Day 180 post transplant
  7-item Likert type scale (from strongly disagree to strongly agree) measures sense of direction and perception of purpose. Scale is 0-7 with 7 = best sense of well-being and 0 = no sense of well-being.
Change in perception and satisfaction with life as assessed by the Meaning in Life Questionnaire and Scale | Pre-BMT and Day 180 post transplant
  Likert-type scale measuring perception of meaning and satisfaction with life (MLQ) Scale is 0-7 with 7 = best sense that life has meaning and 0 = no sense that life has meaning.
Change in personality as measured by the Ten Item Personality Inventory (TIPI) Scale | Pre-BMT and Day 180 post transplant
  7 point Likert-type scale of disagree to agree with various aspects of personality measuring: extraversion, agreeableness, neuroticism, openness, conscientiousness. TIPI scale scoring. Extraversion: 1, 6R; Agreeableness: 2R, 7; Conscientiousness; 3, 8R; Emotional Stability: 4R, 9; Openness to Experiences: 5, 10R. ("R" denotes reverse-scored items)
Change in optimism as assessed by the Life Orientation Scale-Revised | Pre-BMT and Day 180 post transplant
  5 point Likert scale, assessing optimism. 0= strongly disagree; 4 = strongly agree. The total score is from 0 to 24; higher scores indicate more optimism.
Change in perceived loneliness as assessed by the Loneliness Scale | Pre-BMT and Day 180 post transplant
  Revised University of California, Los Angeles (UCLA) Loneliness Scale. Each question is rated on a 4-point scale: 1 = never; 2 = Rarely; 3 = Sometimes 4 = Always. All items are summed to give a total score. Higher scores indicate more loneliness
Change in perceived socio-economic status as assessed by the US socioeconomic questionnaire | Pre-BMT and Day 180 post transplant
  10-rung ladder to assess a participant's perception of participant's status in society. To score this measure, researchers simply note the number of the rung (1-10) on which the respondent placed their "X".
Change in perceived financial strain as assessed by Financial Strain questionnaire | Pre-BMT and Day 180 post transplant
  2 item measure evaluating difficulty and anxiety about money. Higher scores equal higher financial strain.
Change in feeling of community inclusion as assessed by the Social Cohesion Questionnaire | Pre-BMT and Day 180 post transplant
  Participants rate their community by rate of agreement. Response is Agree a lot, a little, do not agree with 3 statements about their community.
Change in feeling of isolation as assessed by the Social Isolation/Engagement Questionnaire | Pre-BMT and Day 180 post transplant
  7-item measure evaluating social isolation, participation and engagement with others. Higher scores= greater sense of isolation.
Change in perceived confidence in spirituality as assessed by the Religion/Spirituality Questionnaire | Pre-BMT and Day 180 post transplant
  5-Item measure for use in epidemiological studies regarding spirituality. Score range from 5-27, with higher scores = more sense of spirituality
Change in feelings of depression as assessed by the Patient Health Questionnaire | Pre-BMT and Day 180 post transplant
  Measures depressive symptoms in the last 2 weeks (PHQ-8)
Change in perceived childhood trauma as assessed by the Adverse Childhood Events (ACE) Scale | Pre-BMT and Day 180 post transplant
  10-item measure to assess childhood abuse and household dysfunction. Response is yes/no. The ACE Scale is scored by summing the number of items for which respondents answered "yes."
Changes in perceived stress as assessed by the Perceived Stress Scale | Pre-BMT and Day 180 post transplant
  5-point Likert scale measures the cognitive appraisal and perceptions of stress in life. Higher score= high level of perceived stress.
Change in bone marrow cell ratios as assessed by Bone Marrow Aspirate | pre-transplant and at Day 180 post-transplant
  aspirate will be collected during standard of care bone marrow biopsies and analyzed using JHU normal reference ranges.
Change in hemoglobin tests. | pre-transplant and then at Day 30, Day 56 and Day 180 post-transplant
  160 mL of blood during evaluations, and 90mL of blood at the day 180 visit. Assessment will be documents using Hopkins normal reference ranges
changes in salivary plasma free cortisol collection | single 24 hour period before BMT and at Day 180 post-transplant
  Saliva collected at home by participants at 4 time points during a single 24 hour period. The mean salivary cortisol concentration is 15.5 +/- 0.8 nmol/L (range, 10.2-27.3) at 0800 h and 3.9 +/- 0.2 nmol/L (range, 2.2-4.1) at 2000 h.
Change in cortisol level | pre-transplant and at Day 180 post-transplant
  This is part of the ACTH Stimulation test to assess the reactivity of hypothalamic-pituitary-adrenal (HPA) axis. Test After the baseline blood draw is taken, 1mcg (low dose) Cosyntropin (synthetic ACTH) will be given intravenously by a research nursing staff followed by serial blood sampling to test for cortisol levels (mcg/dL).
Changes in interleukin (IL)-6 level | pre-transplant and at Day 180 post-transplant
  This is part of the ACTH Stimulation test to assess the reactivity of HPA axis. After the baseline blood draw is taken, 1mcg (low dose) Cosyntropin (synthetic ACTH) will be given intravenously by a research nursing staff followed by serial blood sampling to test for IL-6 levels (pg/ml).
Change in dehydroepiandrosterone (DHEA) level | pre-transplant and at Day 180 post-transplant
  This is part of the ACTH Stimulation test to assess the reactivity of HPA axis. After the baseline blood draw is taken, 1mcg (low dose) Cosyntropin (synthetic ACTH) will be given intravenously by a research nursing staff followed by serial blood sampling to test for DHEA levels (µg/dL).
Change in glucose tolerance as assessed by the Oral Glucose Tolerance Test (OGTT) | pre-transplant and at Day 180 post-transplant
  Participants will fast overnight and then be given the 75 gram glucose oral load followed by blood draws at 0, 30. 60 and 120 minutes. At 120min, below 140mg/dL= normal blood sugar. 200mg/dL or higher= diabetes
Change in heart rate variability as assessed by the "myPatch" Holter monitor | During clinic visits at pre-transplant, Day 30, Day 56 and Day 180
  lightweight digital device that records and stores electrocardiogram (ECG) data on a continuous basis during study visits. A normal resting heart rate for adults ranges from 60 to 100 beats per minute. Generally, a lower heart rate at rest implies more efficient heart function.
Change in attention as assessed by the Flanker Inhibitory Control and Attention Test score | pre-transplant, once a week from Day of transplant to Day 60 and at Day 180 post-transplant
  Measures attention and inhibitory control. Scoring is 0-10. Details and interpretations are available in the NIH toolbox scoring and interpretation guide.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Imus, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT04188678/Prot_SAP_000.pdf